CLINICAL TRIAL: NCT00515411
Title: A Phase II Study of Modified Docetaxel, Cisplatin, and Fluorouracil (mDCF) in Patients With Unresectable or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of Modified Docetaxel, Cisplatin, and Fluorouracil (mDCF) in Unresectable or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry); Roche-Genentech (Industry); City of Hope National Medical Center (Other); Piedmont Hospital Research Institute (Unknown); Medical College of Wisconsin (Other); Queens Health Network (Other); Weill Medical College of Cornell University (Other); Memorial Cancer Institute, Florida (Unknown); University of Pittsburgh (Other); Long Island Jewish Medical Center (Other); Nebraska Cancer Specialists Methodist Estabrook Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-103
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2018-10

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Gastric Cancer
Keywords: gastroesophageal junction; gastric cancer; adenocarcinoma; unresectable gastric cancer; metastatic gastric
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Docetaxel; Leucovorin; Fluorouracil; Cisplatin; pegfilgrastim; Filgrastim; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A, - Modified DCF (Active Comparator): Drug Dose (mg/m2) Schedule
  Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 mg/m2/d daily x 2 days Cisplatin 40 Day 2 OR 3 IVPB (30 min) Arm A is repeated every 2 weeks, and a cycle will be considered 6 weeks (eg 3 treatments).
  Interventions: Drug: Docetaxel, Leucovorin, Fluorouracil, Cisplatin
- ARM B - Parent DCF with G-CSF (Active Comparator): Docetaxel 75 Day 1 IVPB (60 min) Cisplatin 75 Day 1 IVPB (60 min) Fluorouracil 750 IVCI daily x 5 days Neulasta 6 mg subcut on d 8, 9, or 10 or Neupogen 300 or 480 mcg* subcut x 7 d 10-17
  * 300 mcg for weight < 60 kg, 480 mcg for weight > 60 kg
  Interventions: Drug: Docetaxel, Cisplatin, Fluorouracil, Neulasta, or Neupogen
- Arm C - Modifid DCF + Trastuzumab (Active Comparator): Treatment for Her2 Positive Participants
  Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 mg/m2/d daily x 2 days Cisplatin 40 Day 2 OR 3 IVPB (30 min) Trastuzumab Administered on an every 2 week dosing schedule. Initial loading dose of 6 mg/kg over 90 minutes, followed by trastuzumab 4 mg/kg every 2 weeks over 30 minutes.
  Interventions: Drug: Docetaxel, Leukvorin, Flurouracil, Cisplatin, Trastuzumab

INTERVENTIONS:
Drug: Docetaxel, Leucovorin, Fluorouracil, Cisplatin — Drug Dose (mg/m2) Schedule Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 IVCI x 48 hours Cisplatin 40 Day 2 OR 3 IVPB (30 min)
  Arms: Arm A, - Modified DCF
Drug: Docetaxel, Cisplatin, Fluorouracil, Neulasta, or Neupogen — Drug Dose (mg/m2) Schedule Docetaxel 75 Day 1 IVPB (60 min) Cisplatin 75 Day 1 IVPB (60 min) Fluorouracil 750 IVCI daily x 5 days Neulasta 6 mg subcut on d 8, 9, or 10 or Neupogen 300 or 480 mcg* subcut x 7 d 10-17
  * 300 mcg for weight < 60 kg, 480 mcg for weight > 60 kg
  Arm B is repeated every 3 weeks, and a cycle will be considered every 6 weeks (eg 2 treatments). Tumor assessments will be performed following the completion of every cycle for the first 6 cycles, and then every 2 cycles thereafter.
  Arms: ARM B - Parent DCF with G-CSF
Drug: Docetaxel, Leukvorin, Flurouracil, Cisplatin, Trastuzumab — Treatment for Her2 Positive Participants
  Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 mg/m2/d daily x 2 days Cisplatin 40 Day 2 OR 3 IVPB (30 min) Trastuzumab Administered on an every 2 week dosing schedule. Initial loading dose of 6 mg/kg over 90 minutes, followed by trastuzumab 4 mg/kg every 2 weeks over 30 minutes.
  Arms: Arm C - Modifid DCF + Trastuzumab

SUMMARY:
Chemotherapy given together is a standard way to treat your cancer. One standard treatment includes a combination of docetaxel, cisplatin, and fluorouracil. However, the original combination of these three drugs can cause many side effects. This study is being done to find out if these three drugs can be given at lower doses more often, with fewer side effects and still maintain the same benefit as the standard way of giving this three drug combination. If your tumor overexpresses a protein called Her2, you are also eligible to receive trastuzumab with chemotherapy. Trastuzumab is a medicine that has been approved by the US Food and Drug Administration for the treatment of Her2 positive breast cancer. Trastuzumab is now also a standard treatment in combination with chemotherapy for the treatment of Her2 positive stomach cancer. If your tumor is Her2 positive, you would receive the modified administration schedule of docetaxel, cisplatin, and fluorouracil with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or unresectable gastric or gastroesophageal junction (GEJ) adenocarcinoma. GEJ adenocarcinoma may be classified according to Siewert's classification type I, II, or III[43].
* Histological documentation of local recurrence or metastasis is strongly encouraged, unless the risk of such a procedure outweighs the potential benefit of confirming the metastatic disease.
* If no histologic confirmation, then the metastases or recurrence will require documentation by a 2nd radiographic procedure (eg. PET/CT scan or MRI in addition to the CT scan). If the imaging procedure does not confirm recurrent or metastatic disease, biopsy confirmation will be required.
* Patients must have disease that can be evaluated radiographically. This may be measurable disease or non-measurable disease. Measurable disease is defined as that which can be measured in at least one dimension as > 20 mm with conventional techniques, or >10 mm by high resolution imaging. Disease that is identified on radiology studies, but does not meet the criteria for measurable disease, is considered non-measurable.
* Patients may have received no prior chemotherapy for metastatic or unresectable disease. Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and registration. Patients may not have received prior docetaxel or cisplatin.
* Age 18 years or older.
* Karnofsky performance status > than or = to 70% (ECOG performance status 0-1).
* Peripheral neuropathy < than or = to grade 1.
* Hematologic (minimal values):

  * White blood cell count > than or = to 3000/mm3
  * Absolute neutrophil count > than or = to 1500 cells/ mm3
  * Hemoglobin > than or = to 9.0 g/dl
  * Platelet count > than or = to 100,000 / mm3
* Hepatic (minimal values):
* Total bilirubin < or = to 1.5

  * * AST and ALT and Alkaline phosphatase must be within the eligible range. In determining eligibility, the more abnormal of the two values (AST or ALT) should be used. Patients with alkaline phosphatase elevation secondary to the bony metastases rather than liver dysfunction may proceed with treatment on protocol after discussion with the principal investigator.
* Kidney function (minimal values):

  * Serum creatinine < than or = to 1.5 mg/dl - if serum creatinine is 1.2-1.5 mg/dl, the creatinine clearance (either measured or calculated) must be 50 ml/min or greater
* The patient has a PT (INR) < than or = to 1.5 and an PTT < than or = to 3 seconds above the upper limits of normal if the patient is not on anticoagulation. If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:

  * The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW heparin
  * The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Women of childbearing potential have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand informed consent and signing of written informed consent document prior to initiation of protocol therapy.
* Patients must have HER2-positive (FISH+ or IHC 3+) metastatic or unresectable gastric or gastroesophageal junction (GEJ) adenocarcinoma to be eligible for trastuzumab. For the purposes of this protocol, FISH+ is defined as HER2:CEP17 ratio ≥ 2.0. Biopsy samples with cohesive IHC3+ or FISH+ clones are considered HER2 positive irrespective of size, i.e.<10%. FISH+ defined as >2 HER2:CEP17.
* Patients who are receiving trastuzumab must have a left ventricular ejection fraction of ≥ 50%.

Exclusion Criteria:

* Patients who have received previous chemotherapy for the treatment of metastatic or unresectable gastric or GEJ adenocarcinoma are ineligible.
* Patients who have received previous pre- or post-operative chemotherapy or chemoradiation are ineligible if therapy was completed less than 6 months prior to study registration. Patients must have recovered from adverse events from any previous therapy.
* Patients who have received previous docetaxel or cisplatin.
* Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
* Patients with brain or central nervous system metastases, including leptomeningeal disease.
* Pregnant (positive pregnancy test) or breast feeding.
* Serious, non-healing wound, ulcer, or bone fracture.
* Significant cardiac disease as defined as:

unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months

* Evidence of bleeding diathesis or coagulopathy.
* History of a stroke or CVA within 6 months
* Clinically significant peripheral vascular disease.
* Clinically significant hearing loss or ringing in the ears.
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.
* Inability to comply with study and/or follow-up procedures.
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.
* For patients who are Her2 positive and will be treated on the trastuzumab + mDCF cohort, prior trastuzumab treatment is not allowed.
* For patients who are Her2 positive and will be treated on the trastuzumab+mDCF cohort, left ventricular function <50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-10-23 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (15):
  - City of Hope Cancer Center, Duarte, California
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Nebraska Cancer Specialists, Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mondaca S, Margolis M, Sanchez-Vega F, Jonsson P, Riches JC, Ku GY, Hechtman JF, Tuvy Y, Berger MF, Shah MA, Kelsen DP, Ilson DH, Yu K, Goldberg Z, Epstein AS, Desai A, Chung V, Chou JF, Capanu M, Solit DB, Schultz N, Janjigian YY. Phase II study of trastuzumab with modified docetaxel, cisplatin, and 5 fluorouracil in metastatic HER2-positive gastric cancer. Gastric Cancer. 2019 Mar;22(2):355-362. doi: 10.1007/s10120-018-0861-7. Epub 2018 Aug 7. PMID 30088161
- [Derived] Shah MA, Janjigian YY, Stoller R, Shibata S, Kemeny M, Krishnamurthi S, Su YB, Ocean A, Capanu M, Mehrotra B, Ritch P, Henderson C, Kelsen DP. Randomized Multicenter Phase II Study of Modified Docetaxel, Cisplatin, and Fluorouracil (DCF) Versus DCF Plus Growth Factor Support in Patients With Metastatic Gastric Adenocarcinoma: A Study of the US Gastric Cancer Consortium. J Clin Oncol. 2015 Nov 20;33(33):3874-9. doi: 10.1200/JCO.2015.60.7465. PMID 26438119
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A, - Modified DCF: Drug Dose (mg/m2) Schedule
  Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 mg/m2/d daily x 2 days Cisplatin 40 Day 2 OR 3 IVPB (30 min) Arm A is repeated every 2 weeks, and a cycle will be considered 6 weeks (eg 3 treatments).
  Docetaxel, Leucovorin, Fluorouracil, Cisplatin: Drug Dose (mg/m2) Schedule Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 IVCI x 48 hours Cisplatin 40 Day 2 OR 3 IVPB (30 min)
- ARM B - Parent DCF With G-CSF: Docetaxel 75 Day 1 IVPB (60 min) Cisplatin 75 Day 1 IVPB (60 min) Fluorouracil 750 IVCI daily x 5 days Neulasta 6 mg subcut on d 8, 9, or 10 or Neupogen 300 or 480 mcg* subcut x 7 d 10-17 * 300 mcg for weight < 60 kg, 480 mcg for weight > 60 kg
  Docetaxel, Cisplatin, Fluorouracil, Neulasta, or Neupogen: Drug Dose (mg/m2) Schedule Docetaxel 75 Day 1 IVPB (60 min) Cisplatin 75 Day 1 IVPB (60 min) Fluorouracil 750 IVCI daily x 5 days Neulasta 6 mg subcut on d 8, 9, or 10 or Neupogen 300 or 480 mcg* subcut x 7 d 10-17
  * 300 mcg for weight < 60 kg, 480 mcg for weight > 60 kg
  Arm B is repeated every 3 weeks, and a cycle will be considered every 6 weeks (eg 2 treatments). Tumor assessments will be performed following the completion of every cycle for the first 6 cycles, and then every 2 cycles thereafter.
- Arm C - Modified DCF+ Trastuzumab: Treatment for Her2 Positive Participants
  Docetaxel 40 Day 1 IVPB (60 min) Leucovorin 400 Day 1 IVPB (30 min) Fluorouracil 400 IVP day 1 Fluorouracil 1000 mg/m2/d daily x 2 days Cisplatin 40 Day 2 OR 3 IVPB (30 min) Trastuzumab Administered on an every 2 week dosing schedule. Initial loading dose of 6 mg/kg over 90 minutes, followed by trastuzumab 4 mg/kg every 2 weeks over 30 minutes.
Period: Overall Study
Arm/Group | Arm A, - Modified DCF | ARM B - Parent DCF With G-CSF | Arm C - Modified DCF+ Trastuzumab
Started | 54 | 31 | 26
Completed | 54 | 31 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A, - Modified DCF | ARM B - Parent DCF With G-CSF | Arm C - Modified DCF+ Trastuzumab | Total
Number analyzed (Participants) | 54 | 31 | 26 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 23 | 24 | 87
  >=65 years | 14 | 8 | 2 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 3 | 26
  Male | 40 | 22 | 23 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 5 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 45 | 27 | 22 | 94
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 31 | 26 | 111

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Arm A, - Modified DCF | ARM B - Parent DCF With G-CSF | Arm C - Modified DCF+ Trastuzumab
Number analyzed (Participants) | 54 | 31 | 26
percentage of paticipants | 63 [48 to 75] | 53 [34 to 69] | 73 [51 to 86]

2. Secondary Outcome: Overall Survival
Description: Overall survival measured in months
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 43 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A, - Modified DCF | ARM B - Parent DCF With G-CSF | Arm C - Modified DCF+ Trastuzumab
Number analyzed (Participants) | 54 | 31 | 26
months | 18.8 [14.9 to 24.5] | 12.6 [6.7 to 16] | 24.9 [14.4 to 42.5]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm A, - Modified DCF | ARM B - Parent DCF With G-CSF | Arm C - Modified DCF+ Trastuzumab
All-Cause Mortality (participants affected / at risk) | 37/54 | 30/31 | 22/26
Serious Adverse Events (participants affected / at risk) | 26/54 | 23/31 | 13/26
Other Adverse Events (participants affected / at risk) | 26/54 | 23/31 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, - Modified DCF (N=54) | ARM B - Parent DCF With G-CSF (N=31) | Arm C - Modified DCF+ Trastuzumab (N=26)
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1 | 0 | 0
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Cardiac General, other (Cardiac disorders) | 0 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis, infectious (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Creatinine (Investigations) | 0 | 1 | 0
Death not assoc w CTCAE term- Death NOS (General disorders) | 2 | 0 | 2
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 7 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 5
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 0 | 0 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Localized Edema - trunk/genital (General disorders) | 0 | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 | 4 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 0
Fever (in the absence of neutropenia) (General disorders) | 2 | 0 | 5
Fistula, GI- Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal, other (Gastrointestinal disorders) | 3 | 0 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0 | 2
Hematoma (Vascular disorders) | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 2 | 4
Hemorrhage, Stoma (GI) (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, Stomach (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1 | 0 | 1
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 3 | 0 | 0
Inf norm ANC/gr1/2 neut-Catheter-related (Infections and infestations) | 1 | 0 | 0
Inf norm ANC/gr1/2 neut-Urinary(bladder) (Infections and infestations) | 0 | 1 | 1
Inf unknown ANC-Abdomen NOS (Infections and infestations) | 1 | 0 | 0
Infection w/ Gr 3/4 neut, Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0
Infection, other (Infections and infestations) | 2 | 2 | 2
INR (Investigations) | 1 | 0 | 0
Leak, GI- Leak NOS (Gastrointestinal disorders) | 0 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Leukocytes (total WBC) (Investigations) | 2 | 1 | 2
Lymphopenia (Investigations) | 0 | 0 | 1
Metabolic/Lab - Other (specify) (Investigations) | 1 | 0 | 0
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 1 | 1 | 0
Mucositis (func/sympt)- Oral cavity (Gastrointestinal disorders) | 0 | 2 | 0
Muscle weakness - Right-sided (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 9 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 | 1 | 1
Obstruction, GI- Colon (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 2 | 2 | 0
Obstruction, GI- Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 8 | 6 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Cardiac/heart (Cardiac disorders) | 1 | 0 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 0 | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain - Other (specify) (General disorders) | 0 | 0 | 1
Pain - Stomach (Gastrointestinal disorders) | 2 | 0 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Perforation, GI- Cecum (Gastrointestinal disorders) | 0 | 1 | 0
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 4 | 0 | 0
Syncope (fainting) (Nervous system disorders) | 4 | 1 | 2
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 5 | 2 | 1
Ulcer, Esophagus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 10 | 3
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, - Modified DCF (N=54) | ARM B - Parent DCF With G-CSF (N=31) | Arm C - Modified DCF+ Trastuzumab (N=26)
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1 | 0 | 0
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Cardiac General, other (Cardiac disorders) | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis, infectious (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Creatinine (Investigations) | 0 | 1 | 0
Death not assoc w CTCAE term- Death NOS (General disorders) | 2 | 0 | 2
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 7 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 5
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 0 | 0 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Edema: trunk/genital (General disorders) | 0 | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 | 4 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 0
Fever (in the absence of neutropenia) (General disorders) | 2 | 0 | 5
Fistula, GI- Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal, other (Gastrointestinal disorders) | 3 | 0 | 0
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0 | 2
Hematoma (Vascular disorders) | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 2 | 4
Hemorrhage, Stoma (GI) (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, Stomach (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1 | 0 | 1
Hemorrhage/Bleeding, other (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 3 | 0 | 0
Inf norm ANC/gr1/2 neut-Catheter-related (Infections and infestations) | 1 | 0 | 0
Inf norm ANC/gr1/2 neut-Urinary(bladder) (Infections and infestations) | 0 | 1 | 1
Inf unknown ANC-Abdomen NOS (Infections and infestations) | 1 | 0 | 0
Infection w/ Gr 3/4 neut, Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0
Infection, other (Infections and infestations) | 2 | 2 | 2
INR (Investigations) | 1 | 0 | 0
Leak, GI- Leak NOS (Gastrointestinal disorders) | 0 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Leukocytes (total WBC) (Investigations) | 2 | 1 | 2
Lymphopenia (Investigations) | 0 | 0 | 1
Metabolic/Lab - Other (specify) (Investigations) | 1 | 0 | 0
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 1 | 1 | 0
Mucositis (func/sympt)- Oral cavity (Gastrointestinal disorders) | 0 | 2 | 0
Muscle weakness - Right-sided (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 9 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 | 1 | 1
Obstruction, GI- Colon (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 2 | 2 | 0
Obstruction, GI- Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 8 | 6 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Cardiac/heart (Cardiac disorders) | 1 | 0 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 0 | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain - Other (specify) (General disorders) | 0 | 0 | 1
Pain - Stomach (Gastrointestinal disorders) | 2 | 0 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Perforation, GI- Cecum (Gastrointestinal disorders) | 0 | 1 | 0
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 4 | 0 | 0
Syncope (fainting) (Nervous system disorders) | 4 | 1 | 2
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 5 | 2 | 1
Ulcer, Esophagus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 10 | 3
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT00515411/Prot_SAP_000.pdf